CLINICAL TRIAL: NCT05200468
Title: Effect of Intermittent Fasting, Caloric Restriction and Ketogenic Diet on Mitochondrial Function and Gut Microbiota in Subjects With Obesity
Brief Title: Effect of Dietary Restrictions and Ketogenic Diet on Mitochondrial Function and Gut Microbiota in Subjects With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3728
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: dietary restrictions; ketogenic diet; mitochondrial function; gut microbiota
MeSH Terms: conditions — Obesity | interventions — Diet, Ketogenic; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously
Who Masked: Outcomes Assessor
Masking Description: The person who will perform the biochemical determinations, the gut microbiota sequencing and the statistical analysis will be blinded from the intervention group by assigning each patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ketogenic diet (Experimental): Weekly menus will be delivered according to diet with the following macronutrient distribution: 25% protein, 10% carbohydrate, 65% fat. Participants will receive a 30-day food menu guide.
  Interventions: Other: Ketogenic diet
- Caloric restriction diet (Experimental): Weekly menus will be provided according to their usual diet with 500 kcal restriction with the following macronutrient distribution 25-35% protein, 45-55% carbohydrates, 20-30% fat. Participants will receive a 30-day food menu guide.
  Interventions: Other: Caloric restriction diet
- Intermittent fasting 16/8 (Experimental): Calorie-restricted menus will be provided with a 16:8 time-restricted feeding. The feeding window will be 8 hours with a fasting time of 16 hours (04.00 pm- 08.00 am or 05.00 pm - 09.00 am), during the fasting window participants will only be allowed to drink water, unsweetened tea, mineral water and coffee without added sugar. Participants will receive a 30-day food menu guide.
  Interventions: Other: Intermittent fasting 16/8
- habitual diet (No Intervention): Participants will be advised to follow their usual diet until the end of the study.

INTERVENTIONS:
Other: Ketogenic diet — Weekly menus will be delivered according to diet with the following macronutrient distribution: 25% protein, 10% carbohydrate, 65% fat. Participants will receive a 30-day food menu guide.
  Arms: Ketogenic diet
Other: Caloric restriction diet — Weekly menus will be provided according to their usual diet with 500 kcal restriction with the following macronutrient distribution 25-35% protein, 45-55% carbohydrates, 20-30% fat. Participants will receive a 30-day food menu guide.
  Arms: Caloric restriction diet
Other: Intermittent fasting 16/8 — Calorie-restricted menus will be provided with a 16:8 time-restricted feeding. The feeding window will be 8 hours with a fasting time of 16 hours (04.00 pm- 08.00 am or 05.00 pm - 09.00 am), during the fasting window participants will only be allowed to drink water, unsweetened tea, mineral water and coffee without added sugar. Participants will receive a 30-day food menu guide.
  Arms: Intermittent fasting 16/8

SUMMARY:
The benefits of nutritional interventions with dietary restrictions are associated with improvement and preservation of mitochondrial function. Evidence suggests that dietary restrictions, including modifications in caloric intake (caloric restriction), or in the timing of food intake (e.g., intermittent fasting), play an important role in stimulating cell and mitochondrial autophagy, favoring the elimination of old and dysfunctional mitochondria. In addition to the observed effects on mitochondrial function, there is evidence that intermittent fasting, caloric restriction, and the ketogenic diet also generate changes in gut microbiota and microbial metabolite composition. The main aim of this study is to evaluate the effect of intermittent fasting, caloric restriction and ketogenic diet on mitochondrial function determined by respirometry in monocytes, modulated by the gut microbiota in subjects with obesity. An open randomized controlled clinical trial will be conducted with 80 participants divided by a draw in 4 nutritional interventions groups for 1 month, each for 20 participants, then participants will receive 550 mg of rifaximin and will finish the study with the assigned nutritional intervention for another month of follow-up. Knowledge of these dynamics will allow us to explore and understand the relationship between metabolites from the gut microbiota and their effect on mitochondrial function associated with the dietary interventions mentioned above.

DETAILED DESCRIPTION:
The study consists of an open-label randomized controlled clinical trial. Selected subjects will be randomized to one of 4 dietary intervention groups for 1 month with energy intake according to the resting energy expenditure obtained by indirect calorimetry.

The intervention groups will be as follows; a) ketogenic diet, b) caloric restriction diet, c) intermittent fasting diet and, d) usual diet.

1. Ketogenic diet: A dietary recommendation will be given which will be isocaloric according to the resting energy expenditure obtained by indirect calorimetry, containing the following macronutrient distribution: 25% protein, 10% carbohydrates, 65% fat.
2. Caloric restriction diet: A dietary recommendation will be given according to their usual diet, 500 kcal will be restricted, containing the following macronutrient distribution: 25-35% protein, 45-55% carbohydrates, 20-30% fat.
3. Intermittent fasting 16/8: Participants will have the same diet as the participants from the caloric restriction diet group, with the difference that intermittent fasting will be employed, with a time-restricted pattern of 16:8. During 16 hours; for example, from 04.00 pm to 08.00 am or from 05.00 pm to 09.00 am (fasting hours) participants will be fasted and no calories can be eaten or drunk. But participants in the fasting hours can drink water, unsweetened tea, unsweetened coffee and mineral water. In the other 8 hours, participants need to adhere to the energy restriction diet.
4. Usual diet: Participants will not be recommended any diet, participants will be referred to follow their usual diet until the end of the study.

After one month of the assigned intervention, the antibiotic rifaximin will be prescribed to the participants in doses of 550mg, twice a day for 7 days. After the 7 days with the antibiotic, participants will complete another month with the dietary intervention according to the group that the participants were initially randomized.

Participants will be required to complete food logs (2 on weekdays and 1 for weekends) during each week in order to monitor adherence to the dietary plan. For this, a nutritionist will teach them how to complete the food log, where participants must record the type, quantity and place where the food was consumed at each feeding time. Also, 2 phone calls will be made each week to evaluate adherence to treatment. The adherence will be determined with the % of adherence to the dietary treatment as obtained in the analysis of the food logs. Similarly, urine ketone concentration will be determined to measure adherence to the ketogenic diet. A logbook will be provided by the investigator to the participants to record the consumption of the medication, which should be filled out daily by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female.
* Adults between 18 and 60 years of age.
* BMI ≥ 30 and ≤ 50 kg/m2.

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with high blood pressure.
* Patients with acquired diseases secondarily producing obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Patients with gastrointestinal diseases.
* Weight loss > 3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy status.
* Positive smoking.
* Drug treatment:

  * Antihypertensive drugs or treatment
  * Treatment with hypoglycemic agents or insulin and antidiabetic drugs.
  * Treatment with statins, fibrates or other drugs to control dyslipidemia.
  * Use of antibiotics in the three months prior to the study.
  * Use of steroid drugs, chemotherapy, immunosuppressants, or radiation therapy.
  * Anorexigenic or that accelerate weight loss such as sibutramine or orlistat.
  * Supplements with any of the functional foods used in the study.
  * Probiotic, prebiotic or symbiotic supplements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
mitochondrial function | Baseline to 4, 5 and 8 weeks
  Change in mitochondrial function determined by mitochondrial oxygen consumption rate in monocytes

SECONDARY OUTCOMES:
gut microbiota composition | Baseline to 4, 5 and 8 weeks
  Change in microbiota composition determined by alpha and beta diversity analysis to compare the baseline and final microbiota composition between different nutritional interventions in subjects with obesity.
oxidative stress markers | Baseline to 4, 5 and 8 weeks
  Change in markers of oxidative stress determined by levels of malondialdehyde and reactive oxygen species to compare the baseline and final markers of oxidative stress between different nutritional interventions in subjects with obesity.
body composition | Baseline to 4, 5 and 8 weeks
  Change in body composition determined by multifrequency electrical bioimpedance to compare the baseline and final fat mass, lean mass and skeletal muscle mass percentage between different nutritional interventions in subjects with obesity
body weight | Baseline to 4, 5 and 8 weeks
  Change in body weight to compare the baseline and final body weight between different nutritional interventions in subjects with obesity
grip strength | Baseline to 4 and 8 weeks
  Change in grip strength determined by dynamometry to compare the baseline and final grip strength between different nutritional interventions in subjects with obesity.
glucose serum | Baseline to 4 and 8 weeks
  Change in glucose in the serum determined by autoanalyzer to compare the baseline and final concentration of serum glucose between different nutritional interventions in subjects with obesity.
total cholesterol | Baseline to 4 and 8 weeks
  Change in total cholesterol in the serum by autoanalyzer to compare the baseline and final concentration of serum total cholesterol between different nutritional interventions in subjects with obesity
HDL cholesterol | Baseline to 4 and 8 weeks
  Change in HDL cholesterol serum by autoanalyzer to compare the baseline and final concentration of serum HDL-cholesterol between different nutritional interventions in subjects with obesity.
triglycerides | Baseline to 4 and 8 weeks
  Change in triglycerides in the serum by autoanalyzer to compare the baseline and final concentration of serum triglycerides between different nutritional interventions in subjects with obesity.
LDL cholesterol | Baseline to 4 and 8 weeks
  Change in LDL cholesterol in the serum by autoanalyzer to compare the baseline and final concentration of serum LDL cholesterol between different nutritional interventions in subjects with obesity.
leptin | Baseline to 4 and 8 weeks
  Change in leptin concentration in the serum determined by ELISA kit to compare the baseline and final concentration of serum leptin between different nutritional interventions in subjects with obesity.
adiponectin | Baseline to 4 and 8 weeks
  Change in adiponectin concentration in the serum determined by ELISA kit to compare the baseline and final concentration of serum leptin between different nutritional interventions in subjects with obesity.
C-reactive protein | Baseline to 4 and 8 weeks
  Change in C-reactive protein concentration in the serum to compare the baseline and final concentration of serum C- reactive protein between different nutritional interventions in subjects with obesity.
blood pressure | Baseline to 4 and 8 weeks
  Change in systolic and diastolic blood pressure to compare the baseline and final blood pressure between different nutritional interventions in subjects with obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Velazquez Villegas, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts MN, Wallace MA, Tomilov AA, Zhou Z, Marcotte GR, Tran D, Perez G, Gutierrez-Casado E, Koike S, Knotts TA, Imai DM, Griffey SM, Kim K, Hagopian K, McMackin MZ, Haj FG, Baar K, Cortopassi GA, Ramsey JJ, Lopez-Dominguez JA. A Ketogenic Diet Extends Longevity and Healthspan in Adult Mice. Cell Metab. 2017 Sep 5;26(3):539-546.e5. doi: 10.1016/j.cmet.2017.08.005. PMID 28877457
- [Result] Rizza W, Veronese N, Fontana L. What are the roles of calorie restriction and diet quality in promoting healthy longevity? Ageing Res Rev. 2014 Jan;13:38-45. doi: 10.1016/j.arr.2013.11.002. Epub 2013 Nov 27. PMID 24291541
- [Result] Anson RM, Guo Z, de Cabo R, Iyun T, Rios M, Hagepanos A, Ingram DK, Lane MA, Mattson MP. Intermittent fasting dissociates beneficial effects of dietary restriction on glucose metabolism and neuronal resistance to injury from calorie intake. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6216-20. doi: 10.1073/pnas.1035720100. Epub 2003 Apr 30. PMID 12724520
- [Result] Cignarella F, Cantoni C, Ghezzi L, Salter A, Dorsett Y, Chen L, Phillips D, Weinstock GM, Fontana L, Cross AH, Zhou Y, Piccio L. Intermittent Fasting Confers Protection in CNS Autoimmunity by Altering the Gut Microbiota. Cell Metab. 2018 Jun 5;27(6):1222-1235.e6. doi: 10.1016/j.cmet.2018.05.006. PMID 29874567
- [Result] Vidali S, Aminzadeh S, Lambert B, Rutherford T, Sperl W, Kofler B, Feichtinger RG. Mitochondria: The ketogenic diet--A metabolism-based therapy. Int J Biochem Cell Biol. 2015 Jun;63:55-9. doi: 10.1016/j.biocel.2015.01.022. Epub 2015 Feb 7. PMID 25666556
- [Result] Fabbiano S, Suarez-Zamorano N, Chevalier C, Lazarevic V, Kieser S, Rigo D, Leo S, Veyrat-Durebex C, Gaia N, Maresca M, Merkler D, Gomez de Aguero M, Macpherson A, Schrenzel J, Trajkovski M. Functional Gut Microbiota Remodeling Contributes to the Caloric Restriction-Induced Metabolic Improvements. Cell Metab. 2018 Dec 4;28(6):907-921.e7. doi: 10.1016/j.cmet.2018.08.005. Epub 2018 Aug 30. PMID 30174308
- [Result] Lanza IR, Zabielski P, Klaus KA, Morse DM, Heppelmann CJ, Bergen HR 3rd, Dasari S, Walrand S, Short KR, Johnson ML, Robinson MM, Schimke JM, Jakaitis DR, Asmann YW, Sun Z, Nair KS. Chronic caloric restriction preserves mitochondrial function in senescence without increasing mitochondrial biogenesis. Cell Metab. 2012 Dec 5;16(6):777-88. doi: 10.1016/j.cmet.2012.11.003. PMID 23217257
- [Result] Paoli A, Mancin L, Bianco A, Thomas E, Mota JF, Piccini F. Ketogenic Diet and Microbiota: Friends or Enemies? Genes (Basel). 2019 Jul 15;10(7):534. doi: 10.3390/genes10070534. PMID 31311141
- [Result] Hamanaka RB, Chandel NS. Mitochondrial reactive oxygen species regulate cellular signaling and dictate biological outcomes. Trends Biochem Sci. 2010 Sep;35(9):505-13. doi: 10.1016/j.tibs.2010.04.002. Epub 2010 Apr 27. PMID 20430626
- [Result] Ang QY, Alexander M, Newman JC, Tian Y, Cai J, Upadhyay V, Turnbaugh JA, Verdin E, Hall KD, Leibel RL, Ravussin E, Rosenbaum M, Patterson AD, Turnbaugh PJ. Ketogenic Diets Alter the Gut Microbiome Resulting in Decreased Intestinal Th17 Cells. Cell. 2020 Jun 11;181(6):1263-1275.e16. doi: 10.1016/j.cell.2020.04.027. Epub 2020 May 20. PMID 32437658
- [Result] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Derived] Guevara-Cruz M, Hernandez-Gomez KG, Condado-Huerta C, Gonzalez-Salazar LE, Pena-Flores AK, Pichardo-Ontiveros E, Serralde-Zuniga AE, Sanchez-Tapia M, Maya O, Medina-Vera I, Noriega LG, Lopez-Barradas A, Rodriguez-Lima O, Mata I, Olin-Sandoval V, Torres N, Tovar AR, Velazquez-Villegas LA. Intermittent fasting, calorie restriction, and a ketogenic diet improve mitochondrial function by reducing lipopolysaccharide signaling in monocytes during obesity: A randomized clinical trial. Clin Nutr. 2024 Aug;43(8):1914-1928. doi: 10.1016/j.clnu.2024.06.036. Epub 2024 Jul 5. PMID 39003957